CLINICAL TRIAL: NCT03285217
Title: HMB for Denutrition in Patients With Cirrhosis (HEPATIC)
Acronym: HEPATIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Aragones de Ciencias de la Salud (Other Government)
Collaborators: Refbio2: Trans-Pyrenean cooperation network for biomedical research (Unknown)
Responsible Party: Principal Investigator, Jose Miguel Arbones Mainar, Senior Researcher, Instituto Aragones de Ciencias de la Salud
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEPATIC
Record Dates: First submitted 2017-09-11; First posted 2017-09-15 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Sarcopenia; Cirrhosis; Malnutrition
Keywords: HMB
MeSH Terms: conditions — Sarcopenia; Fibrosis; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HMB (Experimental): HMB Group (n=30) will receive received twice a day for 3 months a specialized, nutrient-dense ready-to-drink liquid (Abbott Nutrition) with 350 kcal, 20 g protein, 11 g fat, 44 g carbohydrate, 1.5 g calcium-HMB, 160 IU vitamin D and other essential micronutrients.
  Interventions: Dietary Supplement: Ensure Plus Advance
- Control (Active Comparator): Control Group (n=30) will receive twice a day for 3 months another supplement with similar composition in macro- and micro-nutrients but without HMB
  Interventions: Dietary Supplement: Ensure High Protein

INTERVENTIONS:
Dietary Supplement: Ensure Plus Advance — Supplements, labeled only with the name of the participant and his/her identification number, will be provided to the participants in the Translational Research Unit of the Miguel Servet Hospital. Every 2 weeks, changes in body composition, in particular in fat and muscle, will be assessed by bioelectrical impedance analysis (BIA). Likewise they will be asked about compliance and their diets will be controlled by a nutritionist. Fresh stool samples, urine and blood will be collected pre- and post treatment. An extensive bloodwork will be performed at the Clinical Biochemistry Service at the Miguel Servet Hospital (plasma HMB, total cholesterol, triglycerides, LDL&HDL-cholesterol, free fatty acids, glucose, insulin, β-hydroxybutyrate, hs-CRP, and liver transaminases (AST, ALT, GGT).
  Arms: HMB
Dietary Supplement: Ensure High Protein — Supplements, labeled only with the name of the participant and his/her identification number, will be provided to the participants in the Translational Research Unit of the Miguel Servet Hospital. Every 2 weeks, changes in body composition, in particular in fat and muscle, will be assessed by bioelectrical impedance analysis (BIA). Likewise they will be asked about compliance and their diets will be controlled by a nutritionist. Fresh stool samples, urine and blood will be collected pre- and post treatment. An extensive bloodwork will be performed at the Clinical Biochemistry Service at the Miguel Servet Hospital (plasma HMB, total cholesterol, triglycerides, LDL&HDL-cholesterol, free fatty acids, glucose, insulin, β-hydroxybutyrate, hs-CRP, and liver transaminases (AST, ALT, GGT).
  Arms: Control

SUMMARY:
Cirrhosis is a late stage of hepatic fibrosis caused by many forms of liver diseases and conditions, such as hepatitis and chronic alcoholism. The World Health Organization (WHO) has reported that this condition accounts for 1.8% of all deaths in Europe (170,000 deaths/year).

Patients with cirrhosis are characterized by severe metabolic alterations, which converge in a malnutritional state. Malnutrition encompasses glucose intolerance, chronic inflammation, altered gut microbiota, reduced muscle mass (sarcopenia), as well as loss and dysregulation of adipose tissue (adipopenia). Malnutrition is the most frequent complication that adversely affects the outcomes of cirrhotic patients. Yet, despite its clinical repercussions and potential reversibility, there are no effective therapies because our limited understanding of the mechanisms underlying this altered metabolism.

β-hydroxy β-methylbutyrate (HMB) is a naturally produced substance regarded as safe and effective in preventing muscle loss during chronic diseases. Previous studies have indicated some beneficial effects of HMB itself or its parent metabolite, leucine, on adipose tissue, glucose intolerance, inflammation, and gut microbiota. This study aims to translate those beneficial effects to cirrhotic patients. The investigators hypothesize that HMB can improve cirrhosis-related metabolic abnormalities through its pleiotropic effects. The goals of this study are: i) to perform a randomized clinical trial to evaluate the efficacy of HMB, administered as nutritional supplementation, on clinical symptoms of cirrhosis.

ii) to uncover the precise metabolic pathways that underlie HMB action, with a special focus on muscle, adipose tissue, and gut microbiota.

DETAILED DESCRIPTION:
1. Scientific & technical aspects

State of the art:

Patients with cirrhosis present a chronic inflammatory state and alterations in protein metabolism. These alterations lead to elevated levels of insulin and catecholamines along with the development of glucose intolerance and insulin resistance. The reduced availability of glucose as energy source translates into an accelerated starvation with reduced body fat mass (adipopenia) and loss of skeletal muscle mass (sarcopenia). This catabolic state reduces survival and post-liver transplant outcomes in patients with cirrhosis.

Loss of skeletal muscle mass or sarcopenia is the major component of malnutrition in cirrhosis and occurs in the majority of patients. Impaired ureagenesis and portosystemic shunting provoke skeletal muscle hyperammonemia which induces up-regulation of myostatin and increased autophagy, both of which contribute to sarcopenia.

The adipose tissue (AT) regulates energy homeostasis in the body regardless of the obesity status. Indeed, serum levels of the main adipose-produced cytokines (adipokines) such as leptin, adiponectin, and resistin have been found to be increased in cirrhotic patients as liver function worsens. Evidence demonstrated that adiponectin interacts with the immune/macrophage system and might be of relevance in many liver diseases. Likewise, hyperinsulinemia and increased tumor necrosis factor (TNF) α levels upregulated the adipose resistin gene in rat models of liver cirrhosis.

Recently, growing attention has been targeted to the gut microbiota (GM) in the pathogenesis of gastrointestinal diseases. GM constitutes a symbiotic ecosystem that keeps homeostatic balance within the human body producing a diverse range of compounds that have a major role in regulating the activity of distal organs. Recent studies have shown changes in the relative abundance of microbiota in the stool, colonic mucosa, and saliva of cirrhotic patients. Therefore, modulation of GM arises as a promising tool to prevent and/or to treat the development of these liver disorders.

Clinical guidelines recommend to provide adequate amounts of calories and proteins to cirrhotic patients, either by frequent feeding or via diet supplementation. Consequently, different high caloric diets have been extensively studied. Yet, few studies have shown significant benefit of this type of diets in malnourished cirrhotic patients. Protein supplementation may improve the availability of essential amino acids. However, animal proteins are enriched in aromatic amino acids that are not metabolized by the skeletal muscle and may worsen encephalopathy. Alternatively, modifying the source of nitrogen by using more vegetable protein, less animal protein, and/or branched-chain aminoacids (BCAA) supplementation may help prevent encephalopathy, sarcopenia and adipopenia. Yet, a recently published Cochrane review showed that BCAA did have a beneficial effect on hepatic encephalopathy, but found no effect on mortality, quality of life, or nutritional parameters. This absence of benefit in nutritional parameters might be counter intuitive, as BCAA provide a source of energy to the muscle in addition to being substrates for protein synthesis. The investigators hypothesize that beneficial effects associated to BCAA are, at least partially, mediated by some product/s of their metabolism, likely formed by hepatic synthesis. The cirrhosis-associated liver damage would be hence impeding their synthesis. As consequence, to obtain the expected beneficial outcomes of the BCAA ingestion there should be an increase of the supplemented BCAA or a direct supplementation of the active metabolite/s.

b. Objectives HMB is produced from leucine and is one of its most active metabolites. The majority of HMB production occurs in the liver. Since the mid-1990s, a large body of studies have described that HMB is safe and effective in preventing muscle loss during chronic diseases. Moreover, recent studies have also indicated effects of HMB itself or its parent metabolite, leucine, on adipose tissue differentiation, glucose intolerance, inflammation, gut microbiota, and inflammation reduction. All these beneficial properties make HMB an ideal candidate to supplement the diet of individuals with cirrhosis, a hypothesis that will be tested in the current study. Thus, the specific aim of this proposal is to perform a randomized clinical trial to evaluate the efficacy of HMB, administered as nutritional supplementation, on clinical symptoms of cirrhosis. The study will be performed in adult individuals with cirrhosis. Power analyses based on previously described variations in muscle mass were calculated using R software. The required sample size per group for a power level of 0.9 is estimated to be n = 30,

ELIGIBILITY:
Inclusion Criteria:

1. negative for hepatitis C virus (HCV)&hepatitis B virus (HBV) , or alcohol-caused cirrhosis in stable clinical condition,
2. alcoholic patients must have been abstinent for at least 6 months and be in Child's score of ≤7,
3. no gastrointestinal bleeding for at least 3 months,
4. no clinical, microbiological, or laboratory evidence of infection, renal failure, encephalopathy, malignancy, diabetes mellitus, comorbidities including heart failure or pulmonary disease,
5. No use of medications that affect protein turnover, including corticosteroids and β-blockers.

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in body composition | Baseline, 6 wk, and final (12 wk)
  changes in body composition, in particular in fat and muscle, will be assessed by bioelectrical impedance analysis (BIA)
Liver Status I | Baseline, 6 wk, and final (12 wk)
  Child-Pugh Score
Liver Status II | Baseline, 6 wk, and final (12 wk)
  Liver transaminase enzymes: gamma glutamyl transpeptidase (GGT), aspartate transaminase (AST), and alanine transaminase (ALT) will be combined in a liver functionality score

SECONDARY OUTCOMES:
Nutritional Status I | Baseline, 6 wk, and final (12 wk)
  plasma HMB
Nutritional Status II | Baseline, 6 wk, and final (12 wk)
  Plasma lipids: total cholesterol, triglycerides, LDL&HDL-cholesterol, free fatty acids
Nutritional Status III | Baseline, 6 wk, and final (12 wk)
  Plasma glucose and insulin will be combined to calculate the homeostatic model assessment (HOMA)
Inflammation | Baseline, 6 wk, and final (12 wk)
  C reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Sanz-Paris, MD, Study Director — Hospital Miguel Servet
Locations (1):
- Hospital Universitario Miguel Servet, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Petrides AS, DeFronzo RA. Glucose and insulin metabolism in cirrhosis. J Hepatol. 1989 Jan;8(1):107-14. doi: 10.1016/0168-8278(89)90169-4. PMID 2646365
- [Background] Montano-Loza AJ, Meza-Junco J, Prado CM, Lieffers JR, Baracos VE, Bain VG, Sawyer MB. Muscle wasting is associated with mortality in patients with cirrhosis. Clin Gastroenterol Hepatol. 2012 Feb;10(2):166-73, 173.e1. doi: 10.1016/j.cgh.2011.08.028. Epub 2011 Sep 3. PMID 21893129
- [Background] Qiu J, Thapaliya S, Runkana A, Yang Y, Tsien C, Mohan ML, Narayanan A, Eghtesad B, Mozdziak PE, McDonald C, Stark GR, Welle S, Naga Prasad SV, Dasarathy S. Hyperammonemia in cirrhosis induces transcriptional regulation of myostatin by an NF-kappaB-mediated mechanism. Proc Natl Acad Sci U S A. 2013 Nov 5;110(45):18162-7. doi: 10.1073/pnas.1317049110. Epub 2013 Oct 21. PMID 24145431
- [Background] Floreani A, Variola A, Niro G, Premoli A, Baldo V, Gambino R, Musso G, Cassader M, Bo S, Ferrara F, Caroli D, Rizzotto ER, Durazzo M. Plasma adiponectin levels in primary biliary cirrhosis: a novel perspective for link between hypercholesterolemia and protection against atherosclerosis. Am J Gastroenterol. 2008 Aug;103(8):1959-65. doi: 10.1111/j.1572-0241.2008.01888.x. Epub 2008 Jun 28. PMID 18564121
- [Background] Tilg H, Kaser A, Moschen AR. How to modulate inflammatory cytokines in liver diseases. Liver Int. 2006 Nov;26(9):1029-39. doi: 10.1111/j.1478-3231.2006.01339.x. PMID 17032402
- [Background] Lin SY, Sheu WH, Chen WY, Lee FY, Huang CJ. Stimulated resistin expression in white adipose of rats with bile duct ligation-induced liver cirrhosis: relationship to cirrhotic hyperinsulinemia and increased tumor necrosis factor-alpha. Mol Cell Endocrinol. 2005 Mar 31;232(1-2):1-8. doi: 10.1016/j.mce.2005.01.006. PMID 15737463
- [Background] Betrapally NS, Gillevet PM, Bajaj JS. Gut microbiome and liver disease. Transl Res. 2017 Jan;179:49-59. doi: 10.1016/j.trsl.2016.07.005. Epub 2016 Jul 15. PMID 27477080
- [Background] Plauth M, Cabre E, Riggio O, Assis-Camilo M, Pirlich M, Kondrup J; DGEM (German Society for Nutritional Medicine); Ferenci P, Holm E, Vom Dahl S, Muller MJ, Nolte W; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Liver disease. Clin Nutr. 2006 Apr;25(2):285-94. doi: 10.1016/j.clnu.2006.01.018. Epub 2006 May 16. PMID 16707194
- [Background] Plauth M, Cabre E, Campillo B, Kondrup J, Marchesini G, Schutz T, Shenkin A, Wendon J; ESPEN. ESPEN Guidelines on Parenteral Nutrition: hepatology. Clin Nutr. 2009 Aug;28(4):436-44. doi: 10.1016/j.clnu.2009.04.019. Epub 2009 Jun 11. PMID 19520466
- [Background] Ney M, Vandermeer B, van Zanten SJ, Ma MM, Gramlich L, Tandon P. Meta-analysis: oral or enteral nutritional supplementation in cirrhosis. Aliment Pharmacol Ther. 2013 Apr;37(7):672-9. doi: 10.1111/apt.12252. Epub 2013 Feb 20. PMID 23421379
- [Background] Koretz RL, Avenell A, Lipman TO. Nutritional support for liver disease. Cochrane Database Syst Rev. 2012 May 16;2012(5):CD008344. doi: 10.1002/14651858.CD008344.pub2. PMID 22592729
- [Background] Dasarathy S, Merli M. Sarcopenia from mechanism to diagnosis and treatment in liver disease. J Hepatol. 2016 Dec;65(6):1232-1244. doi: 10.1016/j.jhep.2016.07.040. Epub 2016 Aug 8. PMID 27515775
- [Background] Nguyen DL, Morgan T. Protein restriction in hepatic encephalopathy is appropriate for selected patients: a point of view. Hepatol Int. 2014 Sep 1;8(2):447-51. doi: 10.1007/s12072-013-9497-1. PMID 25525477
- [Background] Gluud LL, Dam G, Les I, Marchesini G, Borre M, Aagaard NK, Vilstrup H. Branched-chain amino acids for people with hepatic encephalopathy. Cochrane Database Syst Rev. 2017 May 18;5(5):CD001939. doi: 10.1002/14651858.CD001939.pub4. PMID 28518283
- [Background] Krebs HA, Lund P. Aspects of the regulation of the metabolism of branched-chain amino acids. Adv Enzyme Regul. 1976;15:375-94. doi: 10.1016/0065-2571(77)90026-7. No abstract available. PMID 19935